CLINICAL TRIAL: NCT02029911
Title: A Multi-Center, Single Arm Clinical Study of the Safety and Efficacy of the AURORA™ Endometrial Ablation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minerva Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP0003
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Menorrhagia Due to Benign Causes
Keywords: Menorrhagia; Excessive uterine bleeding; Endometrial Ablation
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aurora Treatment Arm (Experimental): Endometrial Ablation
  Interventions: Device: Aurora Endometrial Ablation System

INTERVENTIONS:
Device: Aurora Endometrial Ablation System — Ablation of the endometrial lining of the uterus using the Aurora System

SUMMARY:
This is a multi-center, single-arm, non-randomized, prospective clinical study. The clinical study is designed as a non-inferiority study to assess the effectiveness of the Aurora Endometrial Ablation System compared to an objective standard. Safety will be evaluated by determining the number and percentage of subjects who experience one or more of serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory menorrhagia with no definable organic cause
2. Female subject from age 25 to 50 years
3. Uterine sound measurement of 6.0cm to 10.0cm (external os to internal fundus)
4. One of the following criteria:

   A. Documented history of menorrhagia secondary to dysfunctional uterine bleeding (DUB).

   B. If a pictorial blood loss assessment chart (PBLAC) scoring systems is used; a minimum PBLAC score of ≥150 for 1 month prior to study enrollment.
5. Premenopausal at enrollment as determined by FSH measurement ≤ 40 IU/ml
6. Not pregnant and no desire to be pregnant in the future
7. Patient agrees not to use hormonal contraception or any other medical intervention for bleeding during the study
8. Able to provide written informed consent using a form that has been approved by the reviewing IRB/EC
9. Subject agrees to follow-up exams and data collection, including ability to accurately use menstrual diaries for PBLAC analysis.
10. Subject who is literate or demonstrates an understanding on how to use menstrual diaries.

Exclusion Criteria:

1. Pregnancy or subject with a desire to conceive
2. Endometrial hyperplasia as confirmed by histology
3. Presence of active endometritis
4. Active pelvic inflammatory disease
5. Active sexually transmitted disease (STD), at the time of ablation. Note: Treatment of STD documented in the chart serves as sufficient evidence of infection resolution. Patient may be considered for study enrollment.
6. Presence of bacteremia, sepsis, or other active systemic infection
7. Active infection of the genitals, vagina, cervix, uterus or urinary tract at the time of the procedure
8. Known/suspected gynecological malignancy within the past 5 years
9. Known clotting defects or bleeding disorders
10. Untreated/unevaluated cervical dysplasia (except CIN I)
11. Known/suspected abdominal/pelvic cancer
12. Prior uterine surgery (except low segment cesarean section) that interrupts the integrity of the uterine wall (e.g., myomectomy or classical cesarean section)
13. Previous endometrial ablation procedure
14. Currently on medications that could thin the myometrial muscle, such as long-term steroid use (except inhaler or nasal therapy for asthma)
15. Currently on anticoagulants
16. Abnormal or obstructed cavity as confirmed by hysteroscopy or SIS, specifically:

    1. Septate or bicornuate uterus or other congenital malformation of the uterine cavity
    2. Pedunculated or submucosal myomas distorting the uterine cavity
    3. Polyps likely to be the cause of the subject's menorrhagia
    4. Intramural or subserosal myomas that distort the uterine cavity
17. Presence of an intrauterine device (IUD) which the patient is unwilling to have removed at the time of the operative visit
18. Presence of an implantable contraceptive device (e.g. Essure or Adiana).
19. Subject currently on hormonal birth control therapy or unwilling to use a non-hormonal birth control post-ablation (including a Mirena device).
20. Subject who is within 6-weeks post partum.
21. Any general health condition which, in the opinion of the Investigator, could represent an increased risk for the subject
22. Any subject who is currently participating or considers future participation in any other research of an investigational drug or device.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - La Cite Medicale, Québec, Quebec
  - Hôpital Lasalle, Ville Lassalle, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the clinical trial at 3 investigational sites in Canada from June 2011 until October 2011.
Pre-assignment Details: 63 subjects enrolled: 3 subjects excluded based on pre-procedure hysteroscopy screening and did not receive treatment. The remaining 60 subjects completed the study treatment. The protocol ITT population included all subjects in whom treatment was attempted (the experimental device was attempted to be placed).
Period: Overall Study
Arm/Group | Aurora Treatment Arm
Started | 60 (Treatment Attempted)
Treated | 60 (Treatment Completed)
Completed | 60 (Completed 12 Month Follow-up)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects Treated
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 60
PBLAC Score (assessment of menstrual blood loss) [Mean (Standard Deviation); unit: units on a scale] — Pictorial Blood Loss Assessment Chart (PBLAC) is a tool used to assess menstrual blood loss. The PBLAC score takes into account the number of menstrual pads and tampons used as well as amount of saturation. A score of 0 represents no bleeding. Although the PBLAC score does not yield an exact measure of blood loss, it has been found to correlate well with menstrual blood volume. A score greater than 100 is correlated with a blood loss of at least 80 mL.
  units on a scale | 503.0 (412.3)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Menstrual Blood Loss to Normal Levels at 12 Months
Description: Number of subjects in whom menstrual blood loss was reduced to normal or below normal levels at 12 months, as measured by a pictorial blood loss assessment chart (PBLAC) score of <=75.
Time Frame: 12 Months
Population: Protocol Intent-to-treat populations (all subjects in whom the experimental device was attempted to be placed)
Measure: Number; unit: participants
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 60
participants | 58

2. Secondary Outcome: Procedure Time
Description: Procedure Time defined as time from insertion of the Disposable Handpiece to the time of removal.
Time Frame: < 1 hour
Population: Subjects completing treatment
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 60
Minutes | 3.8 (1.3)

3. Post Hoc Outcome: Subjects With Amenorrhea at 12 Months
Description: Amenorrhea at 12 Months- Number of subjects experiencing no menstrual bleeding
Time Frame: 12 Months
Population: Protocol Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Aurora Treatment Arm
Number analyzed (Participants) | 60
participants | 41

ADVERSE EVENTS:
Time Frame: 1 year
Description: All Adverse Events observed during the clinical study, regardless of relationship to the study device or procedure are reported below.
Arm/Group | Aurora Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 53/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aurora Treatment Arm (N=60)
Anesthesia Related (Surgical and medical procedures) | 12 (19)
Vaginal Infection (Reproductive system and breast disorders) | 1 (1)
Bleeding (Reproductive system and breast disorders) | 1 (1)
Pelvic Cramping (non-specific) (Reproductive system and breast disorders) | 47 (57)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Nausea-more than 24 hrs post-treatment (Gastrointestinal disorders) | 2 (2)
Vaginal Discharge (Reproductive system and breast disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4)
Fever more than 24 hrs post-treatment (General disorders) | 2 (2)
Vulvitis (Reproductive system and breast disorders) | 1 (2)
Unpleasant Vaginal Odor (Reproductive system and breast disorders) | 3 (3)
Pruritus Vulvae (Reproductive system and breast disorders) | 1 (1)
Vaginal Burning (Reproductive system and breast disorders) | 1 (1)
Constipaion (Gastrointestinal disorders) | 2 (2)
Superficial Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Vagal Reaction (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Annulus Rectal Condyloma (Infections and infestations) | 1 (1)
Abnormal Pap test- CINII (Reproductive system and breast disorders) | 1 (1)
Dental Ulcer (Gastrointestinal disorders) | 1 (1)
ecchymosis (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No